CLINICAL TRIAL: NCT07344740
Title: Blood Flow Restriction Resistance Exercise and Cardiac Cycle Dynamics
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montclair State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-FY25-26-5034
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Blood flow restriction resistance exercise
  Interventions: Other: Blood flow restriction resistance exercise

INTERVENTIONS:
Other: Blood flow restriction resistance exercise — Blood flow in and out of the limb will be artificially with an occlusion cuff.

SUMMARY:
Blood flow restriction resistance exercise uses partial vascular occlusion of a limb during low weight resistance exercises to stimulate muscle strengthening and growth. This is commonly used during rehabilitation from an injury. Because blood flow in and out of the limbs is decreased, this may have consequences for blood flow through the heart. The purpose of this study will be to test cardiac dynamics during blood flow restriction resistance exercise to determine if cardiac blood flow is impacted. It is hypothesized that both non-BFR exercise and BFR exercise will increase heart rate shortening various cardiac cycle parameters, but BFR exercise will increase the isovolumetric contraction time vs non-BFR exercise due to an increase in total peripheral resistance. It is also hypothesized that BFR exercise will lower early ventricular filling parameters due to lower venous return.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy

Exclusion Criteria:

* Uncontrolled hypertension
* Peripheral vascular disease
* Lymphedema
* Sickle cell anemia
* Heart failure
* Stroke history
* Heart attack history
* Rheumatoid arthritis
* Chronic kidney disease
* Diabetes
* Severe neuropathy
* Any condition that may make blood flow restriction resistance exercise riskier like history of blood clots
* Use of coagulant therapy
* Susceptible to blood clots
* Obesity

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac cycle durations | During the intervention for approximately 10 minutes.
Ventricular filling | During intervention phase for approximately 10 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Montclair State University, Montclair, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No